CLINICAL TRIAL: NCT01648114
Title: A Randomized Controlled Trial of an Antenatal Intervention to Increase Exclusive Breastfeeding
Acronym: ABFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Marie Tarrant, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABFS-1
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breastfeeding; Pregnancy
Keywords: breastfeeding; pregnancy; antenatal; exclusive breastfeeding; education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual outpatient antenatal care consists of routine checking of the maternal and foetal health by either clinic midwives or obstetricians along with health education to promote a healthy pregnancy.
- Antenatal Breastfeeding Intervention (Experimental): Antenatal intervention group will receive usual care plus a 20 to 30-minute one-to-one educational intervention about breastfeeding.
  Interventions: Other: Antenatal Breastfeeding Intervention

INTERVENTIONS:
Other: Antenatal Breastfeeding Intervention — The intervention will include a 20 to 30-minute one-to-one educational talk by a lactation expert explaining the facts of breastfeeding and answering participant questions. The educational intervention will focus on: (1) the importance of exclusive breastfeeding, (2) milk supply/demand and feeding on demand, (3) frequency of feedings, feeding cues, how to know an infant is getting enough milk, (4) avoiding artificial nipples until the infant is nursing well, (5) the importance of a good latch, (5) where to seek breastfeeding help and support, and (7) returning to work and continuing breastfeeding
  Arms: Antenatal Breastfeeding Intervention

SUMMARY:
The investigators will conduct an educational intervention for pregnant women who are planning to breastfeed to promote exclusive breastfeeding and to increase the duration of breastfeeding.

DETAILED DESCRIPTION:
The intervention will include a 20 to 30-minute one-to-one educational talk by a lactation expert explaining the facts of breastfeeding and answering participant questions. The educational intervention will focus on: (1) the importance of exclusive breastfeeding, (2) milk supply/demand and feeding on demand, (3) frequency of feedings, feeding cues, how to know an infant is getting enough milk, (4) avoiding artificial nipples until the infant is nursing well, (5) the importance of a good latch, (5) where to seek breastfeeding help and support, and (7) returning to work and continuing breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnancy,
2. primiparous
3. 18 years of age or older,
4. at least 36 weeks of gestation,
5. Cantonese speaking,
6. Hong Kong resident,
7. no serious medical or obstetrical complications,
8. staying in Hong Kong for at least 6 months after delivery, and
9. intention to breastfeed.

Exclusion Criteria:

Participants will be excluded from the study if they are not entitled to health benefits in Hong Kong (NEP).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Exclusive Breastfeeding Rate | 6 weeks postpartum
  Exclusive breastfeeding rate at 6 weeks postpartum

SECONDARY OUTCOMES:
Median Duration of Breastfeeding | 6 months postpartum
  The median duration of exclusive breastfeeding and the median duration of any breastfeeding
Exclusive Breastfeeding Rate at 3 Months and 6 Months Postpartum | 6 Months Postpartum
  Rate of Exclusive Breastfeeding at 3 Months and 6 Months Postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tarrant, PhD, MPH, RN, Principal Investigator — The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Kwong Wah Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tsan Yuk Hospital, Hong Kong

REFERENCES:
- [Result] Wong KL, Tak Fong DY, Yin Lee IL, Chu S, Tarrant M. Antenatal education to increase exclusive breastfeeding: a randomized controlled trial. Obstet Gynecol. 2014 Nov;124(5):961-968. doi: 10.1097/AOG.0000000000000481. PMID 25437725